CLINICAL TRIAL: NCT01078415
Title: A Prospective, Multi-Center, Clinical Trial Using Irreversible Electroporation (IRE) for the Treatment of Early-Stage Hepatocellular Carcinoma (HCC)
Brief Title: Pilot Study of Irreversible Electroporation (IRE) to Treat Early-Stage Primary Liver Cancer (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-205
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; Hepatocellular Carcinoma; Early Stage; Prospective; Multicenter; Irreversible Electroporation (IRE); Electroporation; Low Energy Direct Current; LEDC; Nonthermal ablation; NTIRE (nonthermal IRE); Ablation; Soft Tissue
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ablation with the NanoKnife Low Energy Direct Current (LEDC) System — 90 pulses of 70 microseconds each in duration will be administered per electrode pair.
  Other Names: System also known as:; * Low Energy Direct Current (LEDC) System; * HVP01 Electroporation System; * NanoKnife LEDC System; * NanoKnife IRE System

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the NanoKnife LEDC System for the treatment of early-stage hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed by positive biopsy or non-invasive criteria,
* not suitable for surgical resection or transplantation,
* have at least one, but less than or equal to 3 tumors,
* of the tumour(s) identified, each tumor must be ≤ 3 cm in diameter,
* Child-Pugh class A,
* Eastern Cooperative Oncology Group (ECOG) score of 0,
* American Society of Anaesthesiologists (ASA) score ≤ 3,
* a prothrombin time ratio > 50%,
* platelet count > 50x109/L,
* ability of patient to stop anticoagulant and anti-platelet therapy for seven days prior to and seven days post NanoKnife procedure,
* are able to comprehend and willing to sign the written informed consent form (ICF),
* have a life expectancy of at least 3 months.

Exclusion Criteria:

* eligible for surgical treatment or transplantation for HCC,
* presence of vascular invasion or extrahepatic metastases,
* received previous treatment for HCC,
* HCC developed on an already transplanted liver,
* cardiac insufficiency, ongoing coronary artery disease or arrhythmia,
* any active implanted device (eg Pacemaker),
* women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* have received treatment with an investigational agent/ procedure within 30 days prior to treatment with the NanoKnife™ LEDC System,
* are in the opinion of the Investigator unable to comply with the visit schedule and protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy as measured by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria by Computed Tomography (CT) or Magnetic Resonance (MR) imaging. | 30 days (+/- 3 days) post treatment

SECONDARY OUTCOMES:
Safety using Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 criteria. | Immediately post treatment to 2 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Lencioni, MD, Principal Investigator — University of Pisa School of Medicine; Jordi Bruix, MD, Principal Investigator — Barcelona Clinic Liver Cancer (BCLC) Group of the University of Barcelona
Locations (6):
- France (2):
  - Hopital Beaujon, Paris
  - L'institut de cancerologie Gustave Roussy, Villejuif, Île-de-France Region
- Universitatsklinikum Magdeburg AoR, Klinik fur Radiologie und Nuklearmedizin, Magdeburg, Germany
- Italy (2):
  - University of Pisa School of Medicine, Pisa, Tuscany
  - Istituto Nazionale Tumori - Fondazione Pascale, Naples
- Barcelona Clinic Liver Cancer Group, Hospital Clinic i Provincial de Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Llovet JM, Burroughs A, Bruix J. Hepatocellular carcinoma. Lancet. 2003 Dec 6;362(9399):1907-17. doi: 10.1016/S0140-6736(03)14964-1. PMID 14667750
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Bruix J, Sherman M, Llovet JM, Beaugrand M, Lencioni R, Burroughs AK, Christensen E, Pagliaro L, Colombo M, Rodes J; EASL Panel of Experts on HCC. Clinical management of hepatocellular carcinoma. Conclusions of the Barcelona-2000 EASL conference. European Association for the Study of the Liver. J Hepatol. 2001 Sep;35(3):421-30. doi: 10.1016/s0168-8278(01)00130-1. No abstract available. PMID 11592607
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Jonas S, Bechstein WO, Steinmuller T, Herrmann M, Radke C, Berg T, Settmacher U, Neuhaus P. Vascular invasion and histopathologic grading determine outcome after liver transplantation for hepatocellular carcinoma in cirrhosis. Hepatology. 2001 May;33(5):1080-6. doi: 10.1053/jhep.2001.23561. PMID 11343235
- [Background] Yao FY, Ferrell L, Bass NM, Watson JJ, Bacchetti P, Venook A, Ascher NL, Roberts JP. Liver transplantation for hepatocellular carcinoma: expansion of the tumor size limits does not adversely impact survival. Hepatology. 2001 Jun;33(6):1394-403. doi: 10.1053/jhep.2001.24563. PMID 11391528
- [Background] Lencioni R, Cioni D, Crocetti L, Franchini C, Pina CD, Lera J, Bartolozzi C. Early-stage hepatocellular carcinoma in patients with cirrhosis: long-term results of percutaneous image-guided radiofrequency ablation. Radiology. 2005 Mar;234(3):961-7. doi: 10.1148/radiol.2343040350. Epub 2005 Jan 21. PMID 15665226
- [Background] Llovet JM, Fuster J, Bruix J. Intention-to-treat analysis of surgical treatment for early hepatocellular carcinoma: resection versus transplantation. Hepatology. 1999 Dec;30(6):1434-40. doi: 10.1002/hep.510300629. PMID 10573522
- [Background] Yao FY, Bass NM, Nikolai B, Davern TJ, Kerlan R, Wu V, Ascher NL, Roberts JP. Liver transplantation for hepatocellular carcinoma: analysis of survival according to the intention-to-treat principle and dropout from the waiting list. Liver Transpl. 2002 Oct;8(10):873-83. doi: 10.1053/jlts.2002.34923. PMID 12360427